CLINICAL TRIAL: NCT03117231
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Knee Osteoarthritis Pain in Elderly Subjects With Defective Endogenous Pain-Inhibitory System: Protocol for a Randomized Clinical Trial
Brief Title: Effects of tDCS in Elderly With Pain Due to Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Daniela Regina Brandão Tavares, Geriatrician, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tavares1
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis, Knee; Chronic Pain
Keywords: osteoarthritis; elderly; musculoskeletal pain; transcranial direct current stimulation
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Osteoarthritis; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Subjects will undergo low-intensity transcranial electrical stimulation for 20 minutes.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Subjects will undergo low-intensity transcranial electrical stimulation for 20 minutes.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Subjects will undergo 15 sessions of tDCS stimulation, 1x per day at 20 minutes per session, of up to 2mA. During active stimulation, the current will be active for the full 20 minutes.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Subjects will undergo 15 sessions of tDCS stimulation, 1x per day at 20 minutes per session, of up to 2mA. However, during sham stimulation (placebo) the current will not be active for the full 20 minutes
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to evaluate if anodal tDCS stimulation over M1 may decrease chronic knee OA pain in elderly subjects with defective CPM. In addition, this trial will help to investigate the role of central sensitization in knee OA and evaluate how tDCS stimulation may affect it.

ELIGIBILITY:
Inclusion Criteria:

* Individuals > 60 years old, of both genders.
* Diagnosis of primary knee osteoarthritis with chronic pain self-reported.
* Be able to sign the informed consent to participate in the study.
* Chronic pain (over the past 6 months) of at least 4 on a 0-10 VAS scale on average.
* Reduction on VAS (visual analogic scale) during CPM (conditioned pain modulation) < 10%

Exclusion Criteria:

* Contraindications to transcranial brain stimulation, i.e. implanted brain medical devices or implanted brain metallic devices.
* Severe acute or chronic decompensated disease.
* Cognitive and behavioral impairment.
* Epilepsy.
* History of fractures in the lower limbs and/or spine in the last 6 months.
* Use of carbamazepine within the past 6 months as self-reported.
* Severe depression (with a score of >30 in the Beck Depression Inventory)
* History of syncope.
* Traumatic brain injury with residual neurological deficits.
* History of alcohol abuse within the past 6 months as self-reported.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Scale | Measured at baseline and up to 60 days after the end of stimulation
  Determine whether anodal transcranial direct current stimulation is effective in reducing pain in subjects with chronic pain due to knee osteoarthritis, as measured by changes in the Brief Pain Inventory (BPI)

SECONDARY OUTCOMES:
Changes in Quality of Life | Measured at baseline, 15, 30 and 60 days after the of stimulation
  The investigators will use the 12-Item Short Form Health Survey (SF-12) to assess changes in quality of life.
Changes in Physical Function as measured through Lequesne Index | Measured at baseline, 15, 30, and 60 days after the end of stimulation
  The investigators will use the Lequesne Index to assess changes in functional capacity.
Changes in Patient Global Assessment | Measured at baseline, 15, 30 and 60 after the end of stimulation
  Modifications in the patient global assessment will be evaluated by measuring changes in the Visual Analogue Scale (VAS).
Changes in Physical Function as measured through Western Ontário and McMaster Universities Osteoarthritis Index | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  The investigators will use the Western Ontário and McMaster Universities Osteoarthritis Index (WOMAC) to assess changes in functional capacity.
Adverse Events | Up to 60 days after the end of stimulation
  Subjects will complete a questionnaire, after each session, to assess potential adverse events of stimulation (headache, neck pain, mood alterations, and seizures) on a 5-point scale.
Changes in Mood | Up to 60 days after the end of stimulation
  The safety of tDCS will be monitored by measuring changes in the Visual Analog Mood Scale.
Changes in cognition | Up to 60 days after the end of stimulation
  The safety of tDCS will be monitored by measuring changes in the MMSE.
One leg standing balance test | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  The investigators will analyse how long time the subject can stay stand on one foot to analise those balance.
Timed Up and Go Test | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  The investigators will measure the walking speed of the subjects.
Changes Pain Pressure Threshold (PPT) | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  Changes in the pain pressure threshold will be analyzed in order to determine whether anodal transcranial direct current stimulation is effective in increasing the pain pressure threshold in subjects with osteoarthritis knee pain.
Changes in mechanical detection threshold as measured through Von-Frey monofilaments | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  Changes in the mechanical detection threshold (MDT) will be measured through calibrated Von-Frey monofilaments in order to determine whether anodal transcranial direct current stimulation is effective in increasing the mechanical detection threshold of subjects with osteoarthritis knee pain.
Changes in mechanical pain threshold as measured through Von-Frey monofilaments | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  Changes in the mechanical pain threshold (MDT) will be measured through calibrated Von-Frey monofilaments in order to determine whether anodal transcranial direct current stimulation is effective in increasing the mechanical pain threshold of subjects with osteoarthritis knee pain.
Descending Noxious Inhibitory Control (DNIC) | Measured at baseline, 15, 30 and 60 days after the end of stimulation
  The investigators will monitore the central modulation of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniela Tavares, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Tavares DRB, Okazaki JEF, Santana MVA, Pinto ACPN, Tutiya KK, Gazoni FM, Pinto CB, Santos FC, Fregni F, Trevisani VFM. Motor cortex transcranial direct current stimulation effects on knee osteoarthritis pain in elderly subjects with dysfunctional descending pain inhibitory system: A randomized controlled trial. Brain Stimul. 2021 May-Jun;14(3):477-487. doi: 10.1016/j.brs.2021.02.018. Epub 2021 Mar 5. PMID 33684598
- [Derived] Tavares DRB, Okazaki JEF, Rocha AP, Santana MVA, Pinto ACPN, Civile VT, Santos FC, Fregni F, Trevisani VFM. Effects of Transcranial Direct Current Stimulation on Knee Osteoarthritis Pain in Elderly Subjects With Defective Endogenous Pain-Inhibitory Systems: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 29;7(10):e11660. doi: 10.2196/11660. PMID 30373731